CLINICAL TRIAL: NCT00746122
Title: Can Emergency Endovascular Aneurysm Repair (eEVAR) Improve the Survival From Ruptured Abdominal Aortic Aneurysm?
Brief Title: Immediate Management of the Patient With Rupture : Open Versus Endovascular Repair
Acronym: IMPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); University of Cambridge (Other); The Leeds Teaching Hospitals NHS Trust (Other); St George's, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTA07/37/64; ISRCTN48334791 (Registry Identifier: ISRCTN registry)
Record Dates: First submitted 2008-09-01; First posted 2008-09-03 (Estimated); Results first posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Conversion to Open Surgery; Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open repair (Other): Immediate Open Surgery
  Interventions: Procedure: Open repair
- Endovascular strategy (Experimental): Endovascular strategy involves immediate computed tomography (CT) and emergency Endovascular aneurysm repair (EVAR), with open repair for patients anatomically unsuitable for EVAR
  Interventions: Procedure: EVAR

INTERVENTIONS:
Procedure: Open repair — Standard treatment of emergency open surgery
  Other Names: open surgical repair; open surgery
  Arms: Open repair
Procedure: EVAR — Emergency endovascular aneurysm repair
  Other Names: Endovascular Aneurysm Repair (EVAR)
  Arms: Endovascular strategy

SUMMARY:
The purpose of this trial is to assess whether a strategy of endovascular repair (if aortic morphology is suitable, open repair if not) versus open repair reduces early mortality for patients with suspected ruptured abdominal aortic aneurysm (AAA).

DETAILED DESCRIPTION:
Rupture of the main blood vessel of the body in the abdomen (ruptured abdominal aortic aneurysm) is fatal in over three-quarters of cases. In the past, those that survive have reached hospital alive and undergone emergency open surgery to repair the aneurysm and stop the bleeding: however, after this major emergency surgery only half the patients leave hospital alive. A newer, less-invasive method of aneurysm repair, endovascular repair, is based on repairing the aneurysm by inserting the repair graft up through one of the arteries in the groin. Endovascular repair has been tested in the elective situation and is associated with a 3-fold reduction in operative mortality versus the standard open surgery. Early work with selected patients has suggested that endovascular repair may be associated with up to a 2-fold reduction in operative mortality and more rapid recovery for ruptured abdominal aortic aneurysms. However, only 55-70% patients are anatomically suitable for endovascular repair.

Therefore, this research aims to determine whether a strategy of preferential emergency endovascular repair reduces both the mortality and cost of ruptured abdominal aortic aneurysm.

Critically ill patients with a clinical diagnosis of ruptured aneurysm will be randomised, in the emergency room, to a strategy of endovascular repair if possible (endovascular first) or to current standard care (immediate transfer to the operating theatre for emergency open surgery). Patients randomised to "endovascular first" will require a specialist radiological examination (computed tomography, CT scan) to assess anatomical suitability and plan for endovascular repair. This will cause a short delay before definitive repair can be commenced. Those patients not suitable for endovascular repair, after CT scan, will be taken for standard open surgery. Patients will be randomised at 16-20 specialist centres in the United Kingdom (UK), who have already attained sufficient experience in using endovascular repair for ruptured aneurysms and can offer a routine service.

The primary outcome measure is 30-day operative mortality, which we hope will improve by 14% with the "endovascular first" strategy (from 47% to 33%). Secondary outcome measures include 24h, in-hospital and 1-year and 3-year mortality, re-interventions associated with the two treatment strategies as well as quality of life, costs and cost-effectiveness.

The research team includes specialists in clinical trials, health economics, statistics, pre-hospital & emergency care, interventional radiology, vascular & endovascular surgery, critical care, aneurysm research and a service user.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of ruptured abdominal aortic aneurysm after review in Accident and Emergency (or other hospital unit).
* Men and women over the age of 50 years will be recruited.

Exclusion Criteria:

* Patients with known connective tissue disorders (eg Marfan syndrome) where endovascular repair may not be beneficial.
* Patients with known previous repair of an abdominal aortic aneurysm, because procedures either open or endovascular are likely to be very complex and there are no guidelines for anatomical restriction to repair.
* Deeply unconscious and moribund patients since the chances of recovery are minimal.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 613 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2013-08-21 (Actual); Study Completion 2016-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ray J. Ashleigh, Principal Investigator — Manchester University NHS Foundation Trust; Simon J. Howell, MRCP(UK) MSc MD, Principal Investigator — Leeds Teaching Hospitals NHS Trust; Ian Chetter, FRCS, Principal Investigator — Hull & East Yorkshire Hospitals NHS Trust; Shane MacSweeney, MA MB BChir MChir FRCSEng, Principal Investigator — Nottingham University Hospitals NHS Trust; Matthew J. Bown, MBChB MD FRCS (Gen Surg), Principal Investigator — University Hospitals, Leicester; Jonathan R Boyle, FRCSEd MD FRCS(Gen), Principal Investigator — Cambridge Vascular Unit, Addenbrooke's Hospital; Meryl Davis, FRCS, Principal Investigator — Royal Free Hampstead NHS Trust; Matthew Thompson, FRCS, Principal Investigator — St George's Healthcare NHS Trust; Colin D Bicknell, FRCS, Principal Investigator — Imperial College NHS Trust; Dynesh Rittoo, MBChB FRCS, Principal Investigator — The Royal Bournemouth & Christchurch Hospitals NHS Foundation Trust; Jonathan Davies, FRCS FRCS(Ed), Principal Investigator — Royal Cornwall Hospitals NHS Trust; Rachel Bell, FRCS, Principal Investigator — Guy's & St Thomas' Hospital; Mike G Wyatt, FRCS, Principal Investigator — The Newcastle upon Tyne Hospitals NHS Trust; Ferdinand Serracino-Inglott, FRCSI, FRCS, Principal Investigator — Manchester Royal Infirmary, Central Manchester University Hospitals NHS Foundation Trust; Paul Bachoo, MBChB FRCS MSc, Principal Investigator — Aberdeen Royal Infirmary; Woolagasen Pillay, FCS(SA), Principal Investigator — Doncaster Royal Infirmary; Syed W Yusuf, FRCS, Principal Investigator — Royal Sussex County Hospital; Paul Walker, Principal Investigator — The James Cook University Hospital , South Tees Hospitals NHS Foundation Trust; Colin Nice, Principal Investigator — Queen Elizabeth Hospital, Gateshead Health NHS Foundation Trust; Andrew Gordon, FRCS, Principal Investigator — Cardiff and Vale University Health Board; Adam Howard, FRCS, Principal Investigator — Colchester General Hospital; Noel Wilson, FRCS MS, Principal Investigator — Kent and Canterbury Hospital; Domenico Valenti, PhD FRCS FEBVS, Principal Investigator — King's College Hospital NHS Trust; David McLain, MBBS, FRCS (Gen Surg), FEBVS, Principal Investigator — Aneurin Bevan Health Board; Patrick Chong, FRCS, Principal Investigator — Frimley Park Hospital NHS Foundation Trust; Raj Bhat,,FRCS(Ed),FRCR, Principal Investigator — NHS Tayside; Luc Dubois, MSc, Principal Investigator — London Health Sciences Centre, University of Western Ontario, Canada; Simon Hobbs, MD, FRCS (Eng), BMedSc, Principal Investigator — The Royal Wolverhampton Hospitals NHS Trust; Stephen Cavanagh, MBChB, MD, FRCS(Gen), Principal Investigator — York Teaching Hospital NHS Foundation Trust; Timothy Rowlands, FRCS (Eng), Principal Investigator — University Hospitals of Derby and Burton NHS Foundation Trust; John Asquith, MRCP, FRCR, Principal Investigator — University Hospital of North Staffordshire
Locations (30):
- London Health Sciences Centre, University of Western Ontario, London, Ontario, Canada
- United Kingdom (29):
  - Royal Cornwall Hospital, Truro, Cornwall
  - University Hospital of Wales, Cardiff and Vale NHS Trust, Cardiff, South Glamorgan
  - The Royal Wolverhampton Hospitals NHS Trust, Wolverhampton, West Midlands
  - Aberdeen Royal Infirmary, NHS Grampian, Aberdeen
  - Royal Bournemouth Hospital, Bournemouth
  - Brighton and Sussex University Hospitals NHS Trust, Brighton
  - Vascular Unit, Addenbrooke's Hospital, Cambridge
  - Kent & Canterbury Hospital, Canterbury
  - Colchester General Hospital, Colchester
  - Royal Derby Hospital, Derby
  - Doncaster and Bassetlaw Hospitals NHS Foundation Trust, Doncaster
  - NHS Tayside, Dundee
  - Frimley Park Hospital NHS Foundation Trust, Frimley
  - Queen Elizabeth Hospital, Gateshead
  - Hull Royal Infirmary, Hull
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Leicester Royal Infirmary, Leicester
  - Royal Free Hampstead NHS Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - St George's Hospital, St George's Healthcare NHS Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Manchester Royal Infirmary, Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - University Hospital of South Manchester, Manchester
  - The James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Royal Gwent Hospital, Newport
  - Queen's Medical Centre, Nottingham
  - The York Hospital, York

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study are/will be available upon request from mjs212@medschl.cam.ac.uk after approval by the Trial Management Committee.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: The data will become available in December 2017 and for the subsequent 3 years.

REFERENCES:
- [Result] IMPROVE Trial Investigators; Powell JT, Sweeting MJ, Thompson MM, Ashleigh R, Bell R, Gomes M, Greenhalgh RM, Grieve R, Heatley F, Hinchliffe RJ, Thompson SG, Ulug P. Endovascular or open repair strategy for ruptured abdominal aortic aneurysm: 30 day outcomes from IMPROVE randomised trial. BMJ. 2014 Jan 13;348:f7661. doi: 10.1136/bmj.f7661. PMID 24418950
- [Result] IMPROVE Trial Investigators. Endovascular strategy or open repair for ruptured abdominal aortic aneurysm: one-year outcomes from the IMPROVE randomized trial. Eur Heart J. 2015 Aug 14;36(31):2061-2069. doi: 10.1093/eurheartj/ehv125. Epub 2015 Apr 7. PMID 25855369
- [Result] Sweeting MJ, Balm R, Desgranges P, Ulug P, Powell JT; Ruptured Aneurysm Trialists. Individual-patient meta-analysis of three randomized trials comparing endovascular versus open repair for ruptured abdominal aortic aneurysm. Br J Surg. 2015 Sep;102(10):1229-39. doi: 10.1002/bjs.9852. Epub 2015 Jun 24. PMID 26104471
- [Result] IMPROVE Trial Investigators. Comparative clinical effectiveness and cost effectiveness of endovascular strategy v open repair for ruptured abdominal aortic aneurysm: three year results of the IMPROVE randomised trial. BMJ. 2017 Nov 14;359:j4859. doi: 10.1136/bmj.j4859. PMID 29138135
- [Derived] Ulug P, Hinchliffe RJ, Sweeting MJ, Gomes M, Thompson MT, Thompson SG, Grieve RJ, Ashleigh R, Greenhalgh RM, Powell JT. Strategy of endovascular versus open repair for patients with clinical diagnosis of ruptured abdominal aortic aneurysm: the IMPROVE RCT. Health Technol Assess. 2018 May;22(31):1-122. doi: 10.3310/hta22310. PMID 29860967
- See also: Improve trial website — https://improvetrial.org/
- Available data/document: Study Protocol — http://www.imperial.ac.uk/department-surgery-cancer/research/surgery/clinical-trials/improve/documents/ — Final protocol version 6.0 dated 28th August 2013

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from 1st September 2009 to 31st July 2013. After 600 recruitment target 13 more patients were randomised before sites could be closed down.
Pre-assignment Details: Exclusions: persons younger than 50 years, prior AAA repair
Groups:
- Endovascular Strategy: Endovascular strategy involves immediate computed tomography (CT) and emergency EVAR, with open repair for patients anatomically unsuitable for EVAR
  EVAR: Emergency endovascular aneurysm repair
Period: Overall Study
Arm/Group | Open Repair | Endovascular Strategy
Started | 297 | 316 (After 600 recruitment target 13 more patients were randomised before sites could be closed down.)
Completed | 297 | 316
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open Repair | Endovascular Strategy | Total
Number analyzed (Participants) | 297 | 316 | 613
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.7 (7.8) | 76.7 (7.4) | 76.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 70 | 133
  Male | 234 | 246 | 480
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 6 | 7 | 13
  United Kingdom | 291 | 309 | 600

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: Mortality, at 3 pre-specified time points
Time Frame: 30 days, 1-year and 3-years from randomisation
Measure: Count of Participants; unit: Participants
Arm/Group | Open Repair | Endovascular Strategy
Number analyzed (Participants) | 297 | 316
Participants
  30-day mortality | 111 | 112
  1-year mortality | 133 | 130
  3-year mortality | 165 | 151

2. Secondary Outcome: Quality-adjusted Life Years (QALYs) to Enable Cost-effectiveness Evaluation
Description: QALYs are a product of length of life and quality of life, since both of these are important to patients. Therefore, it is a measure of the state of health of a person or group in which the benefits, in terms of length of life, are adjusted to reflect the quality of life. One QALY is equal to 1 year of life in perfect health.
  QALYs are calculated by estimating the years of life remaining for a patient following a particular treatment or intervention and weighting each year with a quality-of-life score (on a 0 to 1 scale). It is often measured in terms of the person's ability to carry out the activities of daily life, and freedom from pain and mental disturbance.
Time Frame: 3-years from randomisation
Measure: Mean (Standard Deviation); unit: life-years
Arm/Group | Open Repair | Endovascular Strategy
Number analyzed (Participants) | 297 | 316
life-years | 0.97 (1.02) | 1.14 (1.03)

3. Secondary Outcome: Hospital Costs to Enable Cost-effectiveness Evaluation
Description: Hospital costs to enable cost-effectiveness evaluation in Pounds (£)
Time Frame: 3 years
Measure: Mean (Standard Deviation); unit: GBP (£)
Arm/Group | Open Repair | Endovascular Strategy
Number analyzed (Participants) | 297 | 316
GBP (£) | 19483 (22412) | 16878 (19624)

ADVERSE EVENTS:
Time Frame: During pre-operative Computed Tomography (CT) scan, on days 0 or 1
Description: Death during pre-op CT scan This is an emergency trial where patients die without surgery. This trial compared two types of surgery, endovascular repair and open surgery. The strategy of endovascular repair requires the patient to have a pre-operative CT scan, which may cause a slight delay in reaching the operating theatre. Therefore, the only major adverse event considered during this trial was death during CT scan.
Arm/Group | Open Repair | Endovascular Strategy
All-Cause Mortality (participants affected / at risk) | 297/297 | 316/316
Serious Adverse Events (participants affected / at risk) | 125/297 | 117/316
Other Adverse Events (participants affected / at risk) | 3/243 | 5/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Repair (N=297) | Endovascular Strategy (N=316)
Not discharged from hospital alive (Vascular disorders) | 125 (125) | 117 (117) — Because of the emergency nature of this trial there were no other adverse events monitored
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Repair (N=243) | Endovascular Strategy (N=259)
Major lower limb amputation after aneurysm repair (Vascular disorders) | 3 (3) | 5 (5) — This is only in the patients who underwent emergency repair of AAA rupture, which was limited to 243 in the open repair group and 259 in the endovascular strategy group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes